CLINICAL TRIAL: NCT06190600
Title: Supervised Physical Activity in Young Women With Early Breast Cancer During Neoadjuvant Chemotherpy
Acronym: SPORTNATHy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPORTNATHy
Record Dates: First submitted 2020-01-29; First posted 2024-01-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; physical activity; neoadjuvant chemotherapy; cardiooncology
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — High-Intensity Interval Training; Exercise; Neoadjuvant Therapy; Doxorubicin; Cyclophosphamide; Paclitaxel; Trastuzumab; pertuzumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups. Patients which are set to receive neoadjuvant chemotherapy will be selected. Treatment will be carried out according to 4 x AC regimen (doxorubicin 60 mg/ m2 cyclophosphamide 600 mg/ m2 i.v. every 21 or every 14 days + pegfilgastrim) followed by 12 x paclitaxel 80 mg/ m2 every 7 days and in the case of HER2 positive tumors trastuzumab ± pertuzumab (according to SPC).
  The group in which additional intervention IPA will be ordered, in means of supervised high intensity interval training twice a week. During the course of chemotherapy, the intensity of physical activity will be increasing. Moreover, throughout the entire therapy time, there will be introduced a 45-minute aerobic training session (e.g.: walk, jogging, roller skates, swimming) ones a week. In the control group patients will be asked to independently continue their regular physical activity same as prior to the oncologic treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemotherapy with Standard Supportive Care (Active Comparator): Patients aged 18 to 40 in good physical condition Eastern Cooperative Oncology Group (ECOG) scale 0-1, who are set to receive neoadjuvant chemotherapy will be selected. Criteria for entry into the study include proper liver, kidney and bone marrow function as well as heart ejection fraction of ≥ 50%. Treatment will be carried out according to 4 x AC regimen (doxorubicin 60 mg/ m2 cyclophosphamide 600 mg/ m2 i.v. every 21 or every 14 days + pegfilgastrim) followed by 12 x paclitaxel 80 mg/ m2 every 7 days and in the case of HER2 positive tumors trastuzumab ± pertuzumab (according to SPC).
  Interventions: Drug: neoadjuvant treatment (doxorubicin, cyclophosphamide, paclitaxel, trastuzumab, pertuzumab); Other: Standard Supportive Care
- High Intensity Interval Training (HIIT) (Experimental): The group in which, concurrently with chemotherapy,IPA will be ordered, by means of supervised high intensity interval training twice a week.
  During the course of chemotherapy, the intensity of physical activity will be increasing.
  Interventions: Other: High Intensity Interval Training (HIIT); Drug: neoadjuvant treatment (doxorubicin, cyclophosphamide, paclitaxel, trastuzumab, pertuzumab)

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) — HIIT training twice a week throughout the chemotherapy: treadmill, elliptical, stationary bicycle and indoor rower. The intensity of physical activity will be increasing during consecutive mesocycles. Each training session will begin with a 10-min. wole-body warm-up session at 50-60% hear rate (HR) max. Mesocycle 1 - one month with 4 sets of 1 min. 45 sec. of exercise at a maximal intensity of 75% HR max. Mesocycle 2 with exercises at 80% to 90% HR max divided into 3 periods: 1/ one month, session of 5 sets 1 min. 30 sec. each; 2/ two months, sessions of 5 sets 1 min. 45 sec. each; 3/ two months, sessions of 5 sets 2 min. each. Moreover patients will be instructed to individually perform- a 45-min. aerobic training session (e.g.: walking, jogging, roller skating, swimming) once a week, in patient's own time.
  Other Names: Physical activity
  Arms: High Intensity Interval Training (HIIT)
Drug: neoadjuvant treatment (doxorubicin, cyclophosphamide, paclitaxel, trastuzumab, pertuzumab) — Patients aged 18 to 40 in good physical condition (Eastern Cooperative Oncology Group (ECOG) scale 0-1) who are set to receive neoadjuvant chemotherapy will be selected. Criteria for entry into the study include proper liver, kidney and bone marrow function as well as heart ejection fraction of ≥ 50%. Treatment will be carried out according to 4 x AC regimen (doxorubicin 60 mg/ m2 cyclophosphamide 600 mg/ m2 i.v. every 21 or every 14 days + pegfilgastrim) followed by 12 x paclitaxel 80 mg/ m2 every 7 days and in the case of HER2 positive tumors trastuzumab ± pertuzumab (according to SPC).
  Other Names: chemotherapy
Other: Standard Supportive Care — Patients will be asked to perform 150-300 min. of moderate-intensity aerobic activity or 75-150 min. of vigorous aerobic activity. Each participant will be monitored by an activity watch worn at all times by the patient.
  Other Names: Physical activity
  Arms: Neoadjuvant chemotherapy with Standard Supportive Care

SUMMARY:
The main goal of this study is to assess the impact of supervised intense physical activity (IPA) on outcomes of neoadjuvant chemotherapy in young women with breast cancer (YWBC). In this project standard neoadjuvant chemotherapy will be used concordant with summary of product characteristics (SPC). However during treatment (including days of chemotherapy application) an additional modifier of therapy will be carried out in the form of intense physical activity. This strategy is not recognized in SPC. This project aims to improve the results of breast cancer treatment in young women. According to available data, nowadays this subset of breast cancer patients has worse therapy results in comparison to older women. This is partially because of the different tumor characteristics; young women are more likely to present with human epithelial growth factor receptor 2 (HER2) receptor overexpression or with triple negative breast cancer. In the treatment of YWBC, preoperative chemotherapy is most often the first step. This enables the opportunity to assess the effectiveness of additional interventions in a mode it was never tested before. It is believed that physical activity improves the results of breast cancer treatment, however there are only few reports describing its benefit and role in terms of preoperative chemotherapy.

In the current project, the investigators planned to introduce supervised increased physical activity concurrently with neoadjuvant treatment in YWBC at early stage of disease. The main goal of the study is to assess the effect of physical activity on preoperative chemotherapy outcomes. The change of tumor size after neoadjuvant chemotherapy, as well as the impact on Quality of Life (QoL) and Patients' Reported Outcome (PRO) in described above treatment modality. Secondary endpoints are the following: the pathologic Complete Response (pCR), disease free survival after 3 years (3-yr DFS), overall survival (OS), cardiotoxicity of treatment, the effect of physical activity on tumor microenvironment and Ki67 as well as the impact of increased physical activity on further patients' lifestyle changes.

DETAILED DESCRIPTION:
The main goal of this study is to assess the impact of supervised intense physical activity (IPA) on outcomes of neoadjuvant chemotherapy in young women with breast cancer (YWBC). In this project standard neoadjuvant chemotherapy will be used concordant with summary of product characteristics (SPC). However during treatment (including days of chemotherapy application) an additional modifier of therapy will be carried out in the form of intense physical activity. This strategy is not recognized in SPC. This project aims to improve the results of breast cancer treatment in young women. According to available data, nowadays this subset of breast cancer patients has worse therapy results in comparison to older women. This is partially because of the different tumor characteristics; young women are more likely to present with human epithelial growth factor receptor 2 (HER2) receptor overexpression or with triple negative breast cancer. In the treatment of YWBC preoperative chemotherapy is most often the first step. This enables the opportunity to assess the effectiveness of additional interventions in a mode it was never tested before. It is believed that physical activity improves the results of breast cancer treatment, however there are only few reports describing its benefit and role in terms of preoperative chemotherapy.

In the current project the investigators planned to introduce supervised increased physical activity concurrently with neoadjuvant treatment in YWBC at early stage of disease. The main goal of the study is to assess the effect of physical activity on preoperative chemotherapy outcomes. The change of tumor size after neoadjuvant chemotherapy, as well as the impact on Quality of Life (QoL) and Patients' Reported Outcome (PRO) in described above treatment modality. Secondary endpoints are the following: the pathologic Complete Response (pCR), disease free survival after 3 years (3-yr DFS), overall survival (OS), cardiotoxicity of treatment, the effect of physical activity on tumor microenvironment and Ki67 as well as the impact of increased physical activity on further patients' lifestyle changes. Patients aged 18 to 40 in good physical condition Eastern Cooperative Oncology Group (ECOG) 0-1 who are set to receive neoadjuvant chemotherapy will be selected. Criteria for entry into the study include proper liver, kidney, and bone marrow function as well as heart ejection fraction ≥ 50%. Treatment will be carried out according to 4 x AC regimen (doxorubicin 60 mg/ m2 cyclophosphamide 600 mg/ m2 i.v. every 21 or every 14 days + pegfilgastrim) followed by 12 x paclitaxel 80 mg/ m2 every 7 days and in the case of HER2 positive tumors trastuzumab ± pertuzumab (according to SPC).

After receiving patients' agreement and signing informed consent form, the patient will undergo testing by a multidisciplinary panel of physicians. A cardiological assessment will be completed along with spiroergometry, bone density and anthropometric measurements. The patient will be asked to complete surveys assessing their QoL together with reporting their previous activity level and everyday functioning. Patients will be randomized into two groups - the comparator group undergoing chemotherapy and the intervention group in which additional intervention IPA will be ordered, in means of supervised high intensity interval training twice a week. Modalities of exercise will include: treadmill, elliptical, stationary bicycle and indoor rower. During the course of chemotherapy, the intensity of physical activity will be increasing. Moreover, throughout the entire therapy time, a 45-minute aerobic training session (e.g.: walk, jogging, roller skates, swimming) will be introduced once a week. In the control group, patients will be asked to independently perform their physical activity at an intensity and volume specified in general guidelines: 150-300 min. of moderate-intensity aerobic activity or 75-150 min. of vigorous aerobic activity. Each participant will be monitored at all times by the use of a standard biologic activity recording device.

After the administration of anthracycline, the following procedures will be done: tumor/tumor bed core needle biopsy, mammography, breast ultrasound and cardiological assessment. Following the completion of chemotherapy all testing will be repeated with the exception of bone density measurement and core biopsy. These tests will be repeated one year after surgery. In addition, patients will be assessed for their immune status before and after chemotherapy, as well as one year of observation. When tissue material is available an assessment of the composition of inflammatory infiltrate will be performed using immunohistochemical stainings for immune cell markers. The investigators also planned to preserve material taken from the primary tumor and possible metastasis for molecular analysis (next generation sequencing (NGS), microarrays). The observation will be carried out for 10 years with own resources.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 40 years of age,
* with a known breast cancer, triple - negative or HER2 positive when the tumor size is ≥ 2cm and / or when cancer metastases to axillary lymph nodes or with luminal cancer at tumor size> 3 cm are present,
* qualified for preoperative chemotherapy,
* ECOG 0-1,
* correct left ventricular ejection fraction of at least 50%
* correct results of laboratory tests for bone marrow, liver and kidney function (leukocytes ≥ 3 x 109 / l, neutrocytes ≥ 1.5 x 109 / l, hemoglobin ≥ 9 mg / dl [5.59 mmol / l], platelets ≥ 100 x 109 / l, AST / ALT ≤ 3 x ULN, bilirubin ≤ 1.5 x ULN, creatinine ≤ 1.5 ULN).

Exclusion Criteria:

* diagnosis with cancer other than breast cancer in the last 5 years, except in situ melanoma, in situ cervical cancer, basal cell and squamous cell carcinoma.
* other contraindications for planned systemic treatment: doxorubicin, cyclophosphamide, paclitaxel, trastuzumab, pertuzumab.
* Pregnant and breastfeeding patients.
* Patients infected with HIV, HCV, HBV, after organ transplantation or suffering from an autoimmune disease requiring immunosuppressive treatment. If there are diseases of the musculoskeletal system or other, according to the doctor, preventing the patient from participating in the study or threatening her life and health if the planned intervention is used, the patient should not be included in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in tumor size | 1 year
  Change in tumor size

SECONDARY OUTCOMES:
pathological response | 1 year
  complete pathological response (pCR, pathologic Complete Response)
3-yr DFS | 3 years
  3 years disease-free survival
overall survival | 5 years
  OS - overall survival
Left Ventricle Ejection Fraction (LVEF) | 6 months
  A change in LVEF >10 percentage points, to a value below 50%.
Global Longitudinal Strain (GLS) | 6 months
  A change in GLS >15%.
high-sensitivity troponin | 6 months
  Change above 95 percentile.
BNP | 6 months
  For patients with acute onset dyspnea increase <100 pg/ml, for patients with slow increase in breathlessness increase >35 pg/ml.
Number of steps | 5 years
  Daily number of steps measured throughout the intervention using an activity watch.
Calories burned during physical activity | 5 years
  Measured during physical activity using an activity watch.
Daily calories burned | 5 years
  Measured daily using an activity watch.
Kilometers passed | 5 years
  Measured throughout the intervention using an activity watch.
Time spent actively | 5 years
  Daily number of minutes spent actively measured using an activity watch.
Length of sleep | 5 years
  Daily number of minutes of sleep measured using an activity watch.
Acceptance of illness | 5 years
  Score based on Acceptance of Illness Scale, a single scale with range of points 8-40, with a higher score meaning better acceptance of one's medical condition.
Tumor microenvironment | 1 year
  Assessment of the percentage of immune cells infiltrating the tumor based on immunohistochemical staining of paraffin sections of a tumor. Staining will include the following markers: CD45, CD8, CD4 to assess absolute inflammatory cells, cytotoxic T cells, and helper T cells. The infiltrating cells will be measured as an area occupied by inflammatory cells over total area, and will be expressed as a percentage.
Change in tumor ki67 level | 1 year
  Ki67 will be assessed based on immunohistochemical staining of paraffine section of a tumor. Ki67 index will be measured as a number of ki67-positive cells over the total number of invasive cells, and will be expressed as a percentage.

OTHER OUTCOMES:
PRO-Quality of Life | 5 years
  Score based on the QLQ-BR23 questionnaire which includes the following scales: body image (score range 4-16), sexual functioning (score range 2-8), systemic therapy side effects (score range 7-28), breast symptoms (score range 4-16), arm symptoms (score range 3-12), sexual enjoyment (score range 1-4), future perspectives (score range 1-4), being upset by hair loss (score range 1-4); higher score meaning worse outcome (higher level of symptomatology or lower level of functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Litwiniuk, Prof, Principal Investigator — Wielkopolskie Centrum Onkologii; Joanna Kufel-Grabowska, MD, PhD, Principal Investigator — Wielkopolskie Centrum Onkologii; Maciej Górecki, PT, PhD, Principal Investigator — Wielkopolskie Centrum Onkologii
Locations (1):
- Ewa Tanska, Poznan, Polska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardoso F, Kyriakides S, Ohno S, Penault-Llorca F, Poortmans P, Rubio IT, Zackrisson S, Senkus E; ESMO Guidelines Committee. Early breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2019 Oct 1;30(10):1674. doi: 10.1093/annonc/mdz189. No abstract available. PMID 31236598
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Increasing the dose intensity of chemotherapy by more frequent administration or sequential scheduling: a patient-level meta-analysis of 37 298 women with early breast cancer in 26 randomised trials. Lancet. 2019 Apr 6;393(10179):1440-1452. doi: 10.1016/S0140-6736(18)33137-4. Epub 2019 Feb 8. PMID 30739743
- [Background] Gianni L, Pienkowski T, Im YH, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi GV, Magazzu D, McNally V, Douthwaite H, Ross G, Valagussa P. 5-year analysis of neoadjuvant pertuzumab and trastuzumab in patients with locally advanced, inflammatory, or early-stage HER2-positive breast cancer (NeoSphere): a multicentre, open-label, phase 2 randomised trial. Lancet Oncol. 2016 Jun;17(6):791-800. doi: 10.1016/S1470-2045(16)00163-7. Epub 2016 May 11. PMID 27179402
- [Background] Cardoso F, Harbeck. Breast cancer in young women-a clinical challenge to be addressed in a multidisciplinary setting. Breast Care 2012; 7:193-194
- [Background] Liedtke C, Hess KR, Karn T, Rody A, Kiesel L, Hortobagyi GN, Pusztai L, Gonzalez-Angulo AM. The prognostic impact of age in patients with triple-negative breast cancer. Breast Cancer Res Treat. 2013 Apr;138(2):591-9. doi: 10.1007/s10549-013-2461-x. Epub 2013 Mar 5. PMID 23460246
- [Background] Jones LW, Alfano CM. Exercise-oncology research: past, present, and future. Acta Oncol. 2013 Feb;52(2):195-215. doi: 10.3109/0284186X.2012.742564. Epub 2012 Dec 17. PMID 23244677
- [Background] Bolam KA, Mijwel S, Rundqvist H, Wengstrom Y. Two-year follow-up of the OptiTrain randomised controlled exercise trial. Breast Cancer Res Treat. 2019 Jun;175(3):637-648. doi: 10.1007/s10549-019-05204-0. Epub 2019 Mar 26. PMID 30915663
- [Background] Loughney L, West MA, Kemp GJ, Grocott MP, Jack S. Exercise intervention in people with cancer undergoing neoadjuvant cancer treatment and surgery: A systematic review. Eur J Surg Oncol. 2016 Jan;42(1):28-38. doi: 10.1016/j.ejso.2015.09.027. Epub 2015 Oct 23. PMID 26506862
- [Background] Mugele H, Freitag N, Wilhelmi J, Yang Y, Cheng S, Bloch W, Schumann M. High-intensity interval training in the therapy and aftercare of cancer patients: a systematic review with meta-analysis. J Cancer Surviv. 2019 Apr;13(2):205-223. doi: 10.1007/s11764-019-00743-3. Epub 2019 Feb 26. PMID 30806875
- [Background] West MA, Loughney L, Barben CP, Sripadam R, Kemp GJ, Grocott MP, Jack S. The effects of neoadjuvant chemoradiotherapy on physical fitness and morbidity in rectal cancer surgery patients. Eur J Surg Oncol. 2014 Nov;40(11):1421-8. doi: 10.1016/j.ejso.2014.03.021. Epub 2014 Apr 12. PMID 24784775
- [Background] Betof AS, Lascola CD, Weitzel D, Landon C, Scarbrough PM, Devi GR, Palmer G, Jones LW, Dewhirst MW. Modulation of murine breast tumor vascularity, hypoxia and chemotherapeutic response by exercise. J Natl Cancer Inst. 2015 Mar 16;107(5):djv040. doi: 10.1093/jnci/djv040. Print 2015 May. PMID 25780062
- [Background] Dieli-Conwright CM, Orozco BZ. Exercise after breast cancer treatment: current perspectives. Breast Cancer (Dove Med Press). 2015 Oct 21;7:353-62. doi: 10.2147/BCTT.S82039. eCollection 2015. PMID 26543382
- [Background] Saarto T, Sievanen H, Kellokumpu-Lehtinen P, Nikander R, Vehmanen L, Huovinen R, Kautiainen H, Jarvenpaa S, Penttinen HM, Utriainen M, Jaaskelainen AS, Elme A, Ruohola J, Palva T, Vertio H, Rautalahti M, Fogelholm M, Luoto R, Blomqvist C. Effect of supervised and home exercise training on bone mineral density among breast cancer patients. A 12-month randomised controlled trial. Osteoporos Int. 2012 May;23(5):1601-12. doi: 10.1007/s00198-011-1761-4. Epub 2011 Sep 3. PMID 21892676
- [Background] Rugo HS, Ahles T. The impact of adjuvant therapy for breast cancer on cognitive function: current evidence and directions for research. Semin Oncol. 2003 Dec;30(6):749-62. doi: 10.1053/j.seminoncol.2003.09.008. PMID 14663776
- [Background] Salmon P. Effects of physical exercise on anxiety, depression, and sensitivity to stress: a unifying theory. Clin Psychol Rev. 2001 Feb;21(1):33-61. doi: 10.1016/s0272-7358(99)00032-x. PMID 11148895
- [Background] Furmaniak AC, Menig M, Markes MH. Exercise for women receiving adjuvant therapy for breast cancer. Cochrane Database Syst Rev. 2016 Sep 21;9(9):CD005001. doi: 10.1002/14651858.CD005001.pub3. PMID 27650122
- [Background] Deshmukh SK, Srivastava SK, Poosarla T, Dyess DL, Holliday NP, Singh AP, Singh S. Inflammation, immunosuppressive microenvironment and breast cancer: opportunities for cancer prevention and therapy. Ann Transl Med. 2019 Oct;7(20):593. doi: 10.21037/atm.2019.09.68. PMID 31807574
- [Background] Theriau CF, Connor MK. Voluntary physical activity counteracts the proliferative tumor growth microenvironment created by adipose tissue via high-fat diet feeding in female rats. Physiol Rep. 2017 Jul;5(13):e13325. doi: 10.14814/phy2.13325. PMID 28676553
- [Derived] Gorecki M, Kufel-Grabowska J, Dudek M, Litwiniuk M, Nowak A, Bartczak-Rutkowska A, Straburzynska-Migaj E, Dos J, Marszalek A, Nowaczyk P, Lembryk M, Piotrowski I, Suchorska W, Lesiak M, Marszalek S. A randomized trial on the feasibility of high-intensity interval training during chemotherapy in young breast cancer patients. Sci Rep. 2025 Oct 28;15(1):37591. doi: 10.1038/s41598-025-18377-0. PMID 41152283
- [Derived] Dudek M, Gorecki M, Marszalek S, Kufel-Grabowska J, Litwiniuk M, Nowak A, Bartczak-Rutkowska A, Dos J, Marszalek A, Nowaczyk P, Lembryk M, Piotrowski I, Rosochowicz MA, Suchorska W, Lesiak M, Straburzynska-Migaj E. Supervised high-intensity interval training reduces the negative effect of chemotherapy on cardiorespiratory fitness in young breast cancer women: a randomised controlled study. Eur J Appl Physiol. 2025 Nov;125(11):3141-3154. doi: 10.1007/s00421-025-05822-1. Epub 2025 Jun 5. PMID 40471270